CLINICAL TRIAL: NCT06362772
Title: The Clinical Value of Iodine-125 Seed Implantation in the Treatment of Iodine-refractory Differentiated Thyroid Carcinoma
Brief Title: Clinical Efficacy of 125I Seed Implantation in the Treatment of Refractory Differentiated Thyroid Cancer
Status: Completed | Type: Observational
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MR-36-24-010944
Record Dates: First submitted 2024-04-01; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Thyroid Neoplasms
Keywords: Iodine-125 particles; Brachytherapy; Iodine-refractory differentiated thyroid carcinoma; Thyroid Neoplasms
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Only blood samples were retained to monitor the patient's serum thyroglobulin (Tg), serum anti-thyroglobulin antibody, and thyrotropin (TSH) levels.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 125I seed implantation treatment group: 125I seed implantation treatment group
  Interventions: Radiation: Iodine-125 brachytherapy

INTERVENTIONS:
Radiation: Iodine-125 brachytherapy — In advance of the surgery, patients were informed about their condition, the expected efficacy of 125I seed implantation therapy, alternative treatments such as external beam radiotherapy and chemotherapy, as well as potential side effects and toxic effects. The preoperative evaluation process includes assessments of coagulation function, liver and kidney function, cardiopulmonary function, and local CT scans.
  A collaborative effort between physicians and physicists was undertaken to establish a treatment regimen with a prescription dose ranging from 80 to 120 Gy. The patient accepted the treatment plan and signed an informed consent form. The CT-guided 125I seed implantation procedure was conducted according to the prescribed treatment regimen.
  Efficacy evaluations were conducted at pre-surgery, 1-, 3-, and 5-month post-surgery. The evaluations focused on lesion dimensions, serum Tg, TGAb, TSH levels, pain levels, and adverse reactions.

SUMMARY:
A retrospective analysis was conducted on RAIR-DTC patients who underwent radioactive 125I seed implantation from January 2015 to February 2022 at Jiangxi Cancer Hospital. Prescription dose: 80~120 Gy. All cases were followed up at 1, 3, and 5 months postoperatively to monitor changes in tumor size, serum thyroglobulin (Tg), and serum anti-thyroglobulin antibody levels in thyrotropin-inhibited states, pain scores, and postoperative adverse reactions. The data were processed and analyzed using IBM SPSS 26.0. Pairwise comparisons were conducted using the Wilcoxon signed-rank test, and a p-value of less than 0.05 indicated statistical significance.

DETAILED DESCRIPTION:
Data from RAIR-DTC patients hospitalized at Jiangxi Cancer Hospital from January 2015 to February 2022 were retrospectively collected.

In advance of the surgery, patients were informed about their condition, the expected efficacy of 125I seed implantation therapy, alternative treatments such as external beam radiotherapy and chemotherapy, as well as potential side effects and toxic effects. The preoperative evaluation process includes assessments of coagulation function, liver and kidney function, cardiopulmonary function, and local CT scans.

A collaborative effort between physicians and physicists was undertaken to establish a treatment regimen with a prescription dose ranging from 80 to 120 Gy. The patient accepted the treatment plan and signed an informed consent form. The CT-guided 125I seed implantation procedure was conducted according to the prescribed treatment regimen. Efficacy evaluations were conducted at pre-surgery, 1-, 3-, and 5-month post-surgery. The evaluations focused on lesion dimensions, serum thyroglobulin (Tg), TG antibodies (TGAb), thyroid-stimulating hormone (TSH) levels, pain levels, and adverse reactions.

Lesion size was determined using CT imaging. Lymph nodes were assessed based on their shortest diameter, while other target lesions were evaluated based on their longest diameter. Each measurable lesion underwent an average measurement derived from a minimum of three readings, with all measurements conducted by the same individual to minimize measurement discrepancies.

Response Evaluation Criteria in Solid Tumors (RECIST 1.1) [1] were used to assess treatment response. Use the Visual Analogue Scale to record patients' pain scores. Postoperative adverse reactions, including infection, bleeding, pneumothorax, bone marrow suppression, and seed displacement, were recorded. Radiation injury was graded according to the Radiation Therapy Oncology Group (RTOG) and European Organization for Research and Treatment of Cancer (EORTC) toxicity criteria [2].

The data were analyzed using IBM SPSS 26.0. The count data (n%) and skewed measures [Md (Q1, Q3)] are presented. Group comparisons were conducted using the paired Wilcoxon rank-sum test, with statistical significance set at P < 0.05.

This study was approved by the Ethics Committee of Jiangxi Provincial Cancer Hospital.

ELIGIBILITY:
Inclusion Criteria: Differentiated Thyroid Cancer (DTC) was confirmed by pathology, with local recurrence or distant metastasis of residual thyroid cancer and conforming to any of the following Iodine-Refractory Differentiated Thyroid Cancer (RAIR-DTC) criteria: (1) no uptake of 131I in the initial 131I treatment; (2) loss of iodine uptake capacity in previously functional iodine-avid lesions; (3) disease progression after 131I therapy, including gradual enlargement of the lesion and continuously increasing levels of serum thyroglobulin (Tg).

Exclusion Criteria: Patients with severe physical diseases, such as severe dysfunction of the cardiac, pulmonary, hepatic, or renal systems, poor compliance, inability to tolerate 125I seed implantation, severe acute infectious or chronic infection with acute exacerbation, severe coagulopathy that may lead to serious complications like infection or bleeding, pregnant or lactating women affecting fetal and infant growth and development, patients with cachexia or expected survival of ≤3 Months and patients with positive serum anti-thyroglobulin antibodies (TgAb) that may impact the assessment of treatment efficacy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A retrospective analysis was conducted on Iodine-Refractory Differentiated Thyroid Cancer (RAIR-DTC) patients who underwent radioactive 125I seed implantation from January 2015 to February 2022 at Jiangxi Cancer Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Tumor size | Patients were evaluated preoperatively and at 1, 3, and 5 months postoperatively.
  Lesion size was determined using CT imaging. Lymph nodes were assessed based on their shortest diameter, while other target lesions were evaluated based on their longest diameter. Each measurable lesion underwent an average measurement derived from a minimum of three readings, with all measurements conducted by the same individual to minimize measurement discrepancies. Response Evaluation Criteria in Solid Tumors (RECIST 1.1) were used to assess treatment response[1].
Serological assessment | Patients were evaluated preoperatively and at 1, 3, and 5 months postoperatively.
  Including serum thyroglobulin (Tg) and serum anti-thyroglobulin antibody levels (TgAb) in thyrotropin-inhibited states, as well as tumor markers such as CEA.
Pain score | Patients were evaluated preoperatively and at 1, 3, and 5 months postoperatively.
  Use the Visual Analogue Scale to record patients' pain scores. The scale ranges from 0 to 10 points, with pain increasing incrementally. 0 indicates no pain, 1-3 indicate mild pain that is still tolerable and does not interfere with sleep or normal life, 4-6 indicate moderate pain that interferes with sleep and requires analgesic medication to alleviate it, and 7-10 show intense and intolerable pain that seriously interferes with sleep and diet and requires strong analgesic drugs.
Adverse event | Assess within six months after surgery.
  Postoperative adverse reactions, including infection, bleeding, pneumothorax, bone marrow suppression, and seed displacement, were recorded. Radiation injury was graded according to the Radiation Therapy Oncology Group (RTOG) and European Organization for Research and Treatment of Cancer (EORTC) toxicity criteria [2].

CONTACTS AND LOCATIONS:
Overall Officials: Zhijun Chen, Study Director — Jiangxi Provincial Cancer Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watanabe H, Okada M, Kaji Y, Satouchi M, Sato Y, Yamabe Y, Onaya H, Endo M, Sone M, Arai Y. [New response evaluation criteria in solid tumours-revised RECIST guideline (version 1.1)]. Gan To Kagaku Ryoho. 2009 Dec;36(13):2495-501. Japanese. PMID 20009446
- [Background] Cox JD, Stetz J, Pajak TF. Toxicity criteria of the Radiation Therapy Oncology Group (RTOG) and the European Organization for Research and Treatment of Cancer (EORTC). Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1341-6. doi: 10.1016/0360-3016(95)00060-C. No abstract available. PMID 7713792
- [Derived] Chen Z, Tang X, Tan L, Su Y, Wang W, Wu Z. Efficacy and safety of anlotinib combined with 125I seed implantation for iodine-refractory thyroid cancer. Front Endocrinol (Lausanne). 2025 Aug 22;16:1587412. doi: 10.3389/fendo.2025.1587412. eCollection 2025. PMID 40917344
- [Derived] Wan Q, Tan L, Tang X, Wang W, Su Y, Wu Z, Ke M, Chen Z. The clinical value of iodine-125 seed implantation in the treatment of iodine-refractory differentiated thyroid carcinoma. Front Endocrinol (Lausanne). 2024 Apr 15;15:1327766. doi: 10.3389/fendo.2024.1327766. eCollection 2024. PMID 38686207